CLINICAL TRIAL: NCT02750904
Title: Web-Delivered Acceptance & Commitment Therapy for Smokers With Bipolar Disorder
Acronym: WebQuit Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Palo Alto Veterans Institute for Research (Other); Bedford Research Corporation, Inc. (Other); Jefferson Center, Community Mental Health Clinic (Unknown); VA Central Western Massachusetts Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR File# 8363
Record Dates: First submitted 2016-03-24; First posted 2016-04-26 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Smoking; Bipolar Disorder
Keywords: Smoking Cessation; Acceptance & Commitment Therapy; Cognitive Behavioral Therapy; Bipolar Disorder
MeSH Terms: conditions — Smoking; Bipolar Disorder; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental therapy (Experimental)
  Interventions: Behavioral: Experimental plus Nicotine Replacement Therapy
- Control Therapy (Active Comparator)
  Interventions: Behavioral: Control plus Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Experimental plus Nicotine Replacement Therapy — Behavioral: Experimental plus Nicotine Replacement Therapy will be built to specifically address challenges of smoking cessation for individuals with bipolar disorder.
  Includes four in person and four phone visits.
  Therapy information is withheld to protect the integrity of the study.
  Arms: Experimental therapy
Behavioral: Control plus Nicotine Replacement Therapy — Includes four in-person and four phone visits
  Arms: Control Therapy

SUMMARY:
This purpose of the study is to develop and test a new website to help people who have bipolar disorder quit smoking.

DETAILED DESCRIPTION:
The study consist of two separate phases. Phase I consists of website usability testing. Investigators will collect feedback and incorporate the feedback into our website that is tailored for people with bipolar disorder. In Phase II investigators will be comparing quit rates of two groups both utilizing Nicotine Replacement Therapy and a website.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Daily smoker for the past year, averaging at least 5 cigarettes per day for the past 30 days, with expired-air carbon monoxide (CO) level ≥ 4 ppm
3. Motivated to quit smoking (i.e., endorse plans to quit in the next 30 days at the time of phone pre-screening)
4. Meets lifetime criteria for bipolar I or II disorder, based on DSM-V criteria
5. Willing to be randomly assigned to either treatment group
6. Has at least weekly access to a high-speed Internet connection via a tablet, laptop or desktop computer
7. Willing and able to read in English
8. Is under care of a clinician for the treatment of bipolar disorder
9. Willing to authorize communication with the clinician regarding study participation and clinical deterioration
10. Willing to use the nicotine patch to help quit smoking

Exclusion Criteria:

1. Participating in other smoking cessation interventions
2. Currently using any pharmacotherapies for smoking cessation
3. Previous use of the Smokefree.gov website
4. Meets DSM-V criteria for current mania
5. Meets DSM-V criteria for a current major depressive episode and symptoms are currently severe (Patient Health Questionnaire-9 score > 14)
6. Current psychotic symptoms
7. Psychiatric hospitalization within one month prior to enrollment
8. Current suicidal or homicidal ideation
9. Meets criteria for a DSM-V diagnosis of a moderate or severe substance use disorder in past month prior to enrollment
10. Unstable medical condition
11. Any medical or psychiatric condition that, in the opinion of the investigator, is severe enough to interfere with protocol adherence or ability to benefit from the intervention
12. Any medical conditions that would preclude use of the nicotine patch (e.g., recent myocardial infarction, significant skin disorder, previous severe adverse reaction to nicotine patch, pregnant or breast feeding, assessed with our standard protocol for determining NRT eligibility)
13. Employee or family member of the investigator or study center, or member of the same household as another research participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Recruitment | Week -1 (Visit 0)
  Number approached, screened, eligible, and consented; reasons for ineligibility or refusal
Recruitment | Week 0 (Visit 1)
  Number approached, screened, eligible, and consented; reasons for ineligibility or refusal
Completion of the experimental intervention | Week 10
  Completion of the core treatment program
Retention in study | Week 10
  Percentage of participants in each arm completing outcome assessments at end of treatment visit
Retention in study | Week 14
  Percentage of participants in each arm completing outcome assessments at 1-month follow-up visit
Treatment satisfaction | Week 10
  12 item survey used in our prior work assessing satisfaction with the assigned treatment
Treatment utilization | Week 10
  Server-recorded log-ins to the assigned treatment
Change in acceptance of smoking triggers | Week 10
  Change in acceptance scores between baseline and end of treatment
Change in commitment to quit | Week 10
  Change in commitment scores between baseline and end of treatment
CO-confirmed 7-day point prevalence abstinence from cigarette smoking | Weeks 10
  Preliminary efficacy for smoking cessation
CO-confirmed 7-day point prevalence abstinence from cigarette smoking | Week 14
  Preliminary efficacy for smoking cessation
Change in bipolar disorder symptoms | Week 10
  Change in mania and depression scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Ph.D., Principal Investigator — Fred Hutchinson Cancer Research Institute
Locations (4):
- United States (4):
  - Palo Alto Veterans Institute for Research, Palo Alto, California
  - Jefferson Center for Mental Health, Denver, Colorado
  - Bedford VA Research Corp, Bedford, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: No